CLINICAL TRIAL: NCT00879021
Title: Can Pregabalin Prevent the Development of Neuropathic Pain Following Spinal Cord Injury? A Double-Blind, Randomized, Placebo Controlled Trial.
Brief Title: Study of Pregabalin in the Prevention of Central Neuropathic Pain in Acute Spinal Cord Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding and patients
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Christine Short, MD, FRCPC, FACP, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pregabalin and SCI-Short
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Spinal Cord Trauma; Pain
Keywords: The outcome is to prevent Central Neuropathic Pain; participants will have suffered spinal cord trauma
MeSH Terms: conditions — Spinal Cord Injuries; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin, (other name) Lyrica (Placebo Comparator): Study subjects wil be randomized to either the Pregabalin or Placebo group. There is a 5o ,50 chance of being in either group.
  Interventions: Drug: Lyrica
- pregabalin, drug (Placebo Comparator): study subjects that are randomized to the placebo group will receive matching placebo
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Lyrica — study participants will start will be on 150mg of Pregabalin or placebo capsules by mouth , twice a day.They will be on drug approx. 49 weeks and followed for another 49 weeks after stopping the medication.
  Other Names: Pregablin , also known as Lyrica, an approved drug.
  Arms: Pregabalin, (other name) Lyrica
Drug: matching placebo — 150 mg by mouth ,twice a day for 49 weeks
  Arms: pregabalin, drug

SUMMARY:
This research study will test to see if people who receive pregabalin after their spinal cord injury will develop less nerve damage pain than people who do not receive it.

DETAILED DESCRIPTION:
Pregabalin is one of the few agents that have demonstrated effectiveness in the treatment of central NeP in SCI. Research is now proving that it is possible to prevent the development of pain in certain conditions. Pregabalin has been proven effective in this area with post surgical pain. Therefore, after traumatic SCI there may be a small window of time where we could prevent the development of NeP by administering an agent like Pregabalin.

Objective: To test the hypothesis that pregabalin is an effective treatment in preventing post-spinal cord injury neuropathic pain.

Design: double-blind, placebo controlled, randomized, trial Setting: Spinal cord injury program, neurosurgery and tertiary care rehabilitation center Subjects: 30 patients with acute traumatic spinal cord injury Method: Pregabalin will be offered to patients with acute traumatic spinal cord injury pain in a double blind crossover, placebo control design.

Main Outcome Measures: The primary outcome measures will be the development of Neuropathic Pain and intensity of pain Secondary outcome measures will be Ashworth's Scale for spasticity and ASIA motor and Sensory Scores.

Results: To be determined. Conclusion: To be determined.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 18 years of age or older
* Have suffered a traumatic spinal cord injury (complete or incomplete)
* Be free of Neuropathic pain
* Be in stable medical condition

Exclusion Criteria:

* Pregnant or lactating women: Because we do not know the risks of pregabalin in pregnancy, females of child bearing years must have a negative pregnancy test (performed on screening and subsequent follow up visits) and be using a reliable method of birth control including oral or injectible birth control hormones, barriers, intrauterine devices or tubal ligation, or abstinence throughout the duration of the study.
* Should a female become pregnant while participating in the study she will be un-blinded and, if on pregabalin, she will be weaned from the medication as quickly as is safe and withdrawn from the study. Appropriate follow-up for any pregnancy complications will be conducted.
* Persons with known hypersensitivity to pregabalin or its constituents
* Persons with Neuropathic pain at the time of enrollment
* Persons with a chronic pain diagnoses that may interfere with the evaluation of the presence of Neuropathic pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures will be the development of Neuropathic Pain and intensity of pain . | the trial is 74 weeks in length

SECONDARY OUTCOMES:
Secondary outcome measures will be Ashworth's Scale for spasticity and ASIA motor and Sensory Scores. | trail is 74 weeks in length

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Short, Md FRCPC, Principal Investigator — Capital Health DHA Canada
Locations (1):
- N.S Rehabilitation Center ,Capital Health, Halifax, Nova Scotia, Canada